CLINICAL TRIAL: NCT06673732
Title: Effects of Muscle Energy Technique With and Without Stationary Cycling on Toe Walking With Autism Spectrum Disorder.
Brief Title: Effects of Muscle Energy Technique With and Without Stationary Cycling on Toe Walking With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/Rna Iqbal
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Muscle Energy Technique; Toe-walking; Stationary Cycling
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single( Participant) Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A (n=14) will receive Muscle Energy Technique (MET) combined with stationary Cycling. In the first three days, an initial assessment will be conducted, including Visual Gait Analysis, the Observational Gait Scale, and the Foot Posture Index. From Week 1 to 4, MET will involve the patient contracting for 5-10 seconds while the therapist resists, followed by a rapid 10-second stretch (3-5 repetitions), along with stationary Cycling for 5-10 minutes. A follow-up assessment will occur in Week 4. From Week 5 to 8, the same protocol will continue with 5-8 repetitions and cycling for 10-20 minutes, concluding with a final assessment in Week 8.
  Interventions: Other: Muscle Energy Technique without Stationary Cycling
- Group B (Experimental): Group B (n=14) will undergo Muscle Energy Technique without stationary cycling. In the first 3 days, an initial assessment, including Visual Gait Analysis, Observational Gait Scale, and Foot Posture Index, will be conducted. From Week 1 to 4, the technique involves the patient contracting for 5-10 seconds while the therapist resists, followed by a rapid 10-second stretch (3-5 repetitions). A follow-up assessment will occur in Week 4. From Week 5 to 8, the same process continues with 5-8 repetitions, ending with a final assessment in Week 8.
  Interventions: Other: Muscle Energy Technique with Stationary Bi-Cyclying

INTERVENTIONS:
Other: Muscle Energy Technique with Stationary Bi-Cyclying — MET for post-isometric relaxation of the Achilles, calf, quads, hamstrings, and ankle, position each muscle at resistance, just short of pain. The patient contracts (10-20% effort) for 5-10 seconds while the therapist resists. After relaxing and exhaling, the therapist gently stretches the muscle to the new barrier. Repeat this process 2-3 times, gradually increasing the stretch with each repetition.
  For PFS MET of the Achilles tendon, calf, quads, hamstrings, and ankle, contract the muscle maximally for 5-10 seconds while the therapist resists. Afterward, the muscle is relaxed, and the therapist quickly stretches it to the new barrier, holding for 10 seconds. Following a 20-second rest, repeat the process 3-5 times. For Reciprocal Inhibition MET, the muscle is placed mid-range, the patient pushes against resistance, then relaxes while the therapist stretches the muscle. This is repeated 3-5 times. Stationary cycling complements the routine.
  Arms: Group B
Other: Muscle Energy Technique without Stationary Cycling — MET for post-isometric relaxation of the Achilles, calf, quads, hamstrings, and ankle, position each muscle at resistance, just short of pain. The patient contracts (10-20% effort) for 5-10 seconds while the therapist resists. After relaxing and exhaling, the therapist gently stretches the muscle to the new barrier. Repeat this process 2-3 times, gradually increasing the stretch with each repetition. Post FS MET of the Achilles tendon, calf, quads, hamstrings, and ankle, contract the muscle maximally for 5-10 seconds while the therapist resists. Afterward, the muscle is relaxed, and the therapist quickly stretches it to the new barrier, holding for 10 seconds. Following a 20-second rest, repeat the process 3-5 times. For Reciprocal Inhibition MET, the muscle is placed mid-range, the patient pushes against resistance, then relaxes while the therapist stretches the muscle. This is repeated 3-5 times without Stationary Cycling
  Arms: Group A

SUMMARY:
In Autism spectrum disorder (ASD) is a developmental disability caused by differences in the brain. People with ASD often have problems with social communication and interaction, and restricted or repetitive behaviors or interests. People with ASD may also have different ways of learning, moving, or paying attention. The Aim of this thesis is Effects of Muscle Energy Technique with and without Stationary Cycling on toe walking children with Autism Spectrum Disorder This study seeks to explore whether the synergistic application of these interventions can provide a more comprehensive and effective approach in managing the debilitating symptoms associated with toe walking in Autistic children.

DETAILED DESCRIPTION:
. The study's sample size will be 26 participants. Inclusion criteria for this study will be: Diagnosed Autistic between ages 4-10 years, Diagnosed Autistic Children, Treatment was given to each of the participants for 3 days a week and for 8 weeks. Inclusion criteria were all gender with the age group of 4-10 years, participants diagnosed cases of Autism spectrum disease with Toe Walking and their exclusion criteria were suspected but undiagnosed cases of ASD, the presence of any limb deformities , autistic children with MR, and unwillingness of participant or parents to be a part of the study. An RCT included 26 diagnosed autistic children as per inclusion criteria the subjects were divided into two groups, i.e., group A and B, the group A was given MET with Stationary bicycling whereas Group B was given MET without Stationary Bi-Cycling participants were clinically examined. Dynamometer, foot posture Index, Observational Gait Scale, and Parent report of percentage of time toe walking,

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosed Autism .
* Aged between 4 to 10 years.
* Autistic children with Toe-Walking
* Regular for follow-up
* Both Gender included

Exclusion Criteria:

* Children with Comorbidities .
* Children with mild cognitive dysfunction
* Children less then 4 year or older than 10 years..
* Autistic Children with limb deformity
* Autistic Children with Mental Retardation.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-01-07 (Estimated); Study Completion 2025-01-07 (Estimated)

PRIMARY OUTCOMES:
Observational Gait Scale | 8 weeks
  Observational Gait Scale An Assessment/observational gait exam is the Observational Gait Scale (OGS). The OGS is primarily used to rate gait metrics using a structured scale from video recordings It focuses on the knee joint and foot position during mid-stance. . In routine clinical practice, observational gait evaluation is regarded as a more economical option to IGA. The purpose of this paper is to evaluate the validity and reliability of the various pediatric gait analysis techniques by doing a thorough evaluation and comparing them to IGA.(20) The OGS score's validity was assessed by contrasting it with the 3-DGA. For knee and foot posture in mid-stance, first foot contact, and heel rise, the OGS was shown to have satisfactory interrater and intrarater reliability with weighted kappas (wk) ranging from 0.53 to 0.91 (intrarater) and 0.43 to 0.86 (interrater).

SECONDARY OUTCOMES:
foot Posture Index | 5-10 minutes
  The Foot Posture Index (FPI) assesses foot alignment using six criteria, including talar head position, arch height, and heel alignment. Each criterion is scored from -2 to +2, indicating levels of supination (negative) or pronation (positive). The total score classifies the foot as supinated, neutral, or pronated. It's a useful tool for identifying foot posture and potential biomechanical issues.
Foot Dynamometer: | 8 weeks
  A foot dynamometer is a device used to measure the strength and force exerted by the foot muscles. It assesses grip strength, particularly in the toes, and is often used in sports science and rehabilitation to evaluate foot function, stability, and recovery progress. The dynamometer provides objective data on muscle force, which helps guide therapy for foot injuries or biomechanical issues

CONTACTS AND LOCATIONS:
Overall Officials: Rna Mohammad Iqbal, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lord C, Brugha TS, Charman T, Cusack J, Dumas G, Frazier T, Jones EJH, Jones RM, Pickles A, State MW, Taylor JL, Veenstra-VanderWeele J. Autism spectrum disorder. Nat Rev Dis Primers. 2020 Jan 16;6(1):5. doi: 10.1038/s41572-019-0138-4. PMID 31949163